CLINICAL TRIAL: NCT06234735
Title: A Personalized Physical Activity Intervention and Behavioral Change in Lung Cancer Patients: RETOS Pilot Study
Brief Title: Physical Activity Behavioral Change Intervention in Lung Cancer
Acronym: RETOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Collaborators: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1399
Record Dates: First submitted 2023-09-08; First posted 2024-01-31 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer; Sedentary Behavior; Fatigue
Keywords: Physical activity; Community; Physiotherapy
MeSH Terms: conditions — Lung Neoplasms; Sedentary Behavior; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator and the professional who will do the statistical analyses, will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will follow the conventional protocol established by the Catalan Institute of Oncology (ICO) for the treatment of lung cancer. In addition, physical activity guidelines will be recommended with the aim of encouraging patients to lead a more active life that helps them improve their physical capabilities. The research team will meet individually with participants in the control group and inform them about the importance of physical activity, motivating them to practice regularly.
  Interventions: Behavioral: Conventional intervention
- Experimental Group (Experimental): Motivational interviews will be used to help identify individual motivations, barriers, and preferences towards physical activity (PA). Objectives and personalized exercise regimens (e.g. walking, cycling, nordic walking) with a person-centered approach. Patients will engage in a minimum of 3 PA sessions/week (45min each) for 6 months, reporting via a phone app. Weekly patient-reported outcome measures (PROMs) will track progress. The first 3 months involve group sessions for instruction and correction; the last 3 months include one monthly in-person session combining resistance and aerobic training, with a duration of 1.5 hours. To drive behavior change, personalized weekly challenges will be presented.
  Interventions: Behavioral: Physical activity in the community

INTERVENTIONS:
Behavioral: Physical activity in the community — Supervised and guided PA sessions in the community setting using public resources such as parks, sports facilities, etc.
  Arms: Experimental Group
Behavioral: Conventional intervention — Conventional protocol for lung cancer and PA recommendations.
  Arms: Control Group

SUMMARY:
Patients with lung cancer have poor physical activity and increased sedentary behavior, with the presence of high levels of fatigue.

A randomized controlled trial will be carried out to compare usual care versus a personalized exercise program in the community, in order to explore the changes on physical activity and sedentary behavior and its impact on cancer-related fatigue.

DETAILED DESCRIPTION:
Patients with lung cancer are characterized by having low levels of physical activity (PA) and high sedentary behavior (SB), with direct impact on their quality of life, complications and survival. Previous studies have observed that PA programs have high dropout rates and are not very sustainable over time, making it necessary to incorporate models that consider the preferences and possibilities of patients.

Objectives: To compare the effects on PA levels and SB of a 6-month personalized program vs. conventional care, in community-dwelling lung cancer survivors.

Methods: Controlled and randomized pilot study, with intervention and control group, pilot study. 40 non-small cell lung cancer survivors (18 to 70 years old) will be included. The control group will receive the usual recommendations regarding an active and healthy lifestyle. The intervention group will follow a personalized PA and behavior change program in the community, supervised by a physiotherapist expert in therapeutic exercise.

PA and SB measurements will be carried out using accelerometry and self-reported questionnaires. As secondary variables, functional capacity, lung function, dyspnea and fatigue, as well as quality of life will be measured. A motivational interview will be conducted to personalize the intervention considering clinical characteristics, treatment, motivation and preferences. The intervention will be re-evaluated and adapted monthly, considering the results reported weekly.

Through covariance analysis, the levels of PA and SB, among other factors, measured at the beginning and at the end of the intervention will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of non-small cell lung cancer who are candidates for radical and/or metastatic treatment
* ages between 18 and 70
* ability to answer questionnaires in Spanish
* who have accepted participation and signed the informed consent

Exclusion Criteria:

* participants with a life expectancy of less than 6 months
* patients with levels of physical activity greater than 240 metabolic equivalents (MET) METs/day
* patients who have a contraindication to exercise
* patients with dementia or spatial disorientation or behavioral disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | 7 consecutive days, before and after intervention (6 months)
  Level of daily physical activity measured with accelerometry. Accelerometry will be worn by patients for 7 consecutive days and will measure the time in minutes spent in low (1.6 - <3 METs), moderate (3.0 - <6.0 METs) and vigorous (⩾6 METs) physical activities.
Sedentarism | Before and after intervention (6 months)
  Weekly sedentary behavior measured with the Sedentary Behaviour Questionnaire (SBQ). The SBQ measures the time in minutes spent in 9 different sedentary activities during a week, differentiating working days and week-ends. The score is the separately sum of the hours per day for week days and week-end days. A higher score is indicative of longer time spent in sitting and therefore an indication of higher sedentarism.

SECONDARY OUTCOMES:
Walking distance | Before and after intervention (6 months)
  The six-minute walking test (6MWT) will be used to determine walking distance, in meters (m), covered during six minutes. A 30-meter indoor corridor will be used and patients will be encouraged to walk as much as possible during that time.
1-minute Sit-to-Stand test | Before and after intervention (6 months)
  Number of sit-to- stand repetitions done in 1 minute (STS-1m). A 46-cm high chair will be used.
Pulmonary function | Before and after intervention (6 months)
  Forced spirometry following the American Thoracic Society (ATS) and European Respiratory Society (ERS) recommendations. The following variables will be obtained from the spirometry: forced vital capacity (FVC, in percentage (%); forced expiratory volume first second (FEV1), in percentage (%).
Dyspnea | Before and after intervention (6 months), and once a week during intervention.
  The modified Medical Research Council (mMRC) scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 meters or after a few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing.
Cancer Quality of Life Questionnaire | Before and after intervention (6 months).
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire and Lung Cancer Module (EORTC QLQ-LC13) is a quality of life questionnaire specific for cancer. It is designed to measure cancer patients' physical, psychological and social functions. The questionnaire consists of multi-item scales and single items. Items are scored 1 to 4 and a higher score indicates more symptom burden.
Fatigue | Before and after intervention (6 months), and once a week during intervention.
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 13-item questionnaire specific for cancer patients to assess the intensity and impact of fatigue on daily life in the last 7 days. Respondents use a 5-point Likert-type scale ranging from 0 (not at all) to 4 (very much). Responses are added to create a total score (possible range 0 to 52). Higher scores reflect higher levels of fatigue experimented by the patient.
Adherence | Once a week during intervention period (6 months).
  The total number of completed PA sessions followed by patients during the intervention period in relation to the total number of planified sessions.
IPAQ short form | Before and after intervention (6 months).
  The International Physical Activity Questionnaire (IPAQ), will provide the subjective perception of time spent in different levels of PA. It is calculated in metabolic equivalent (MET)-minutes per week, calculated as the MET intensity multiplied by the minutes for each activity over the last 7 days and the time spent sitting. Classified with low (1.6 - <3 METs), moderate (3.0 - <6.0 METs) and vigorous (⩾6 METs) physical activities.
Hand grip test | Before and after intervention (6 months).
  The hand grip force will be measured by digital dynamometry. The measure will be in kilograms (kg).
Calf circumference | Before and after intervention (6 months).
  The calf circumference will be assessed with a measuring tape in centimeters (cm) looking for the maximal perimeter. This measure is to assess the skeletal muscle status.
Bioimpedance | Before and after intervention (6 months).
  Bioimpedance (BIA) will be used to estimate body fat and muscle mass. Fat free mass (FFM) in percentage (%), fat mas (FM) in percentage (%), total body water (TBW) in percentage (%), and body cell mass (BCM) in percentage (%), will be measured.
Sleep quality | Before and after intervention (6 months), and once a week during intervention period (6 months).
  The Pittsburgh sleep quality index (PSQI) assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. The PSQI questions are rated from 0 = no difficulty to 3 = severe difficulty, generating scores that correspond to the domains of the scale. The scores range from 0 to 21 and a score >5 be considered as a significant sleep disturbance.

OTHER OUTCOMES:
Daily dyspnea | Before and after each physical activity session, minimum 3 sessions per week, during the intervention period (6 months).
  During the 6-month intervention period, dyspnea perception will be measured before and immediately after each PA session with the modified Borg scale. This is a 0 to 10 scale, that shows the maximum dyspnea, 10, and 0 no dyspnea at all.
Steps per day | Once a week during intervention (6 months)
  During the 6-month intervention period, number of daily steps measured with App pedometer will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Teixido, PhD, Study Chair — University Ramon Llull
Locations (1):
- Blanquerna Health Science Faculty, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No